CLINICAL TRIAL: NCT03092453
Title: Mature Dendritic Cell Vaccination Against Mutated Antigens in Patients With Advanced Melanoma
Brief Title: Dendritic Cell Vaccination in Patients With Advanced Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 17616, 826433; 17616 (Other: Abramson Cancer Center)
Record Dates: First submitted 2017-03-07; First posted 2017-03-28 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vaccines; Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mature dendritic cell (DC) vaccine (Experimental): Mature DC 7.5-15 million/peptide given day 1, every six weeks for 2 doses followed by standard of care anti PD-1 therapy
  Interventions: Biological: Mature dendritic cell (DC) vaccine; Drug: Cyclophosphamide 300mg/m^2; Drug: Pembrolizumab

INTERVENTIONS:
Biological: Mature dendritic cell (DC) vaccine — Mature DC 7.5-15 million/peptide followed by 2 booster every six weeks of 1-5 million/peptide followed by standard of care anti PD-1 therapy.
Drug: Cyclophosphamide 300mg/m^2 — administered prior to subject's first DC dose
Drug: Pembrolizumab — administered 7-8 weeks after subject's last DC dose

SUMMARY:
The purpose of this study is to investigate a method of using dendritic cells (a kind of white blood cell) as a vaccine to stimulate your own immune system to react to your melanoma cells.

DETAILED DESCRIPTION:
This is a single arm open label trial that will assess the safety and tolerability of mature dendritic cell (mDC3/8) vaccine (primer and booster) in subjects with stage III and stage IV melanoma, followed by treatment with pembrolizumab (anti-PD-1 therapy).

Eligible patients that provide written informed consent will undergo apheresis to collect blood mononuclear cells for vaccine production approximately 1 week prior to vaccine infusion. Each study subject will receive cyclophosphamide 300mg/m^2 intravenously or by mouth 3 to 4 days prior to the vaccine dose, to deplete regulatory T cells. For each vaccine dose, all subjects will receive autologous dendritic cells pulsed with melanoma tumor-specific peptides. On Day 1, the subject will receive the primer vaccine dose; this will be followed by two booster vaccine doses at 6 weeks apart. Peripheral blood will be taken weekly to monitor the immune response to each peptide by tetramer assay. Re-staging will occur after the 3rd vaccine dose, along with tumor biopsy and second apheresis. Anti PD-1 therapy (standard of care) will commence 7-8 weeks after the subject's last dendritic cell vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage III and stage IV M1a/M1b/M1c melanoma. Measurable disease is not required for enrollment eligibility and patients with completely resected disease are permitted.
* Male or female patients age greater than or equal to 18 years
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Required initial laboratory values (performed within 14 days prior to eligibility confirmation by physician-investigator):

  * WBC (white blood cells) >3,000/mm3
  * Hg (hemoglobin) greater than or equal to 9.0 gm/dl
  * Platelets >75,000/mm3
  * Serum Bilirubin < 2.0 mg/dl
  * Serum Creatinine < 2.0 mg/dl
* Subjects of reproductive potential must agree to use a medically accepted birth control method during the trial and for at least two months following the trial.
* Provide written informed consent.

Exclusion Criteria:

* Prior treatment with more than one line of cytotoxic chemotherapy; prior treatment with one line of cytotoxic chemotherapy is permitted. Prior treatment with targeted therapy (such as ipilimumab, anti-PD1, or BRAF + MEK inhibitor combination) is permitted.
* Active untreated CNS (central nervous system) metastasis
* Active infection
* Prior malignancy (except non-melanoma skin cancer) within 3 years
* Pregnant or nursing (lactating) women
* Concurrent treatment with high-dose systemic corticosteroids; local (inhaled or topical) steroids are permitted
* Known allergy to eggs
* Prior history of uveitis or autoimmune inflammatory eye disease
* Known positivity for hepatitis B antibody, hepatitis C antibody, or HIV antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald P Linette, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mature Dendritic Cell (DC) Vaccine
Started | 5
Completed | 3
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mature Dendritic Cell (DC) Vaccine
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Immune Response Measuring Increased Numbers of Peptide Specific T Cells as Calculated by the Tetramer Assay.
Description: Immune response measuring increased numbers of peptide specific T cells as calculated by the tetramer assay. The numbers of Peptide Specific T Cells are reported as the percent of CD8+ T cells that were p/HLA multimer positive for each antigen.
Time Frame: Screening through week 21
Population: Antigens for each subject may be different. Outcomes were not tested past week 21.
Measure: Number; unit: percent of CD8+ T cells
Groups:
- Subject 1; Subject 2; Subject 3; Subject 4: Mature DC 7.5-15 million/peptide given day 1, every six weeks for 2 doses followed by standard of care anti PD-1 therapy
  Mature dendritic cell (DC) vaccine: Mature DC 7.5-15 million/peptide followed by 2 booster every six weeks of 1-5 million/peptide followed by standard of care anti PD-1 therapy.
  Cyclophosphamide 300mg/m^2: administered prior to subject's first DC dose
  Pembrolizumab: administered 7-8 weeks after subject's last DC dose
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4
Number analyzed (Participants) | 1 | 1 | 1 | 1
percent of CD8+ T cells
  Antigen A3-1, screening: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-1, screening | 0 |  | 0 | 0
  Antigen A3-2, screening: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-2, screening | 0 |  | 0 | 0
  Antigen A3-3, screening: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-3, screening | 0 |  | 0 | 0
  Antigen A3-4, screening: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-4, screening | 0 |  | 0 | 0
  Antigen A3-5, screening: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-5, screening | 0 |  | 0 | 0
  Antigen A3-6, screening: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-6, screening | 0 |  | 0 | 0
  Antigen A3-7, screening: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-7, screening | 0 |  | 0 |
  Antigen B8-1, screening: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-1, screening | 0 |  |  |
  Antigen B8-3, screening: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-3, screening | 0.26 |  |  |
  Antigen B8-4, screening: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-4, screening | 0 |  |  |
  Antigen B8-5, screening: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-5, screening | 0 |  |  |
  Antigen A3-1, Day 1: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-1, Day 1 | 0 |  | 0 | 0
  Antigen A3-2, Day 1: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-2, Day 1 | 0 |  | 0 | 0
  Antigen A3-3, Day 1: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-3, Day 1 | 0 |  | 0 | 0
  Antigen A3-4, Day 1: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-4, Day 1 | 0 |  | 0 | 0
  Antigen A3-5, Day 1: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-5, Day 1 | 0 |  | 0 | 0
  Antigen A3-6, Day 1: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-6, Day 1 | 0 |  | 0 | 0
  Antigen A3-7, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen A3-7, Day 1 | 0 |  |  |
  Antigen B8-1, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-1, Day 1 | 0.4 |  |  |
  Antigen B8-3, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-3, Day 1 | 0.48 |  |  |
  Antigen B8-4, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-4, Day 1 | 0 |  |  |
  Antigen B8-5, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-5, Day 1 | 0 |  |  |
  Antigen A3-1, wk 14-15: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-1, wk 14-15 | 0 |  | 0 | 0.86
  Antigen A3-2, wk 14-15: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-2, wk 14-15 | 0 |  | 0 | 2.66
  Antigen A3-3, wk 14-15: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-3, wk 14-15 | 0 |  | 0 | 0
  Antigen A3-4, wk 14-15: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-4, wk 14-15 | 0 |  | 0 | 4.01
  Antigen A3-5, wk 14-15: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-5, wk 14-15 | 0 |  | 0 | 0
  Antigen A3-6, wk 14-15: number analyzed (Participants) | 1 | 0 | 1 | 1
  Antigen A3-6, wk 14-15 | 0 |  | 2.4 | 0
  Antigen A3-7, wk 14-15: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen A3-7, wk 14-15 | 0 |  |  |
  Antigen B8-1, wk 14-15: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-1, wk 14-15 | 0.32 |  |  |
  Antigen B8-3, wk 14-15: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-3, wk 14-15 | 5.68 |  |  |
  Antigen B8-4, wk 14-15: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-4, wk 14-15 | 0 |  |  |
  Antigen B8-5, wk 14-15: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-5, wk 14-15 | 0 |  |  |
  Antigen A3-1, wk 17: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-1, wk 17 | 0 |  | 0 |
  Antigen A3-2, wk 17: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-2, wk 17 | 0 |  | 0 |
  Antigen A3-3, wk 17: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-3, wk 17 | 0 |  | 0 |
  Antigen A3-4, wk 17: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-4, wk 17 | 0 |  | 0 |
  Antigen A3-5, wk 17: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-5, wk 17 | 0 |  | 0 |
  Antigen A3-6, wk 17: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-6, wk 17 | 0 |  | 0 |
  Antigen A3-7, wk 17: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen A3-7, wk 17 | 0 |  |  |
  Antigen B8-1, wk 17: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-1, wk 17 | 0.5 |  |  |
  Antigen B8-3, wk 17: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-3, wk 17 | 1.81 |  |  |
  Antigen B8-4, wk 17: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-4, wk 17 | 0 |  |  |
  Antigen B8-5, wk 17: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-5, wk 17 | 0 |  |  |
  Antigen A3-1, wk 19: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-1, wk 19 | 0 |  | 0 |
  Antigen A3-2, wk 19: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-2, wk 19 | 0 |  | 0 |
  Antigen A3-3, wk 19: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-3, wk 19 | 0 |  | 0 |
  Antigen A3-4, wk 19: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-4, wk 19 | 0 |  | 0 |
  Antigen A3-5, wk 19: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-5, wk 19 | 0 |  | 0 |
  Antigen A3-6, wk 19: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-6, wk 19 | 0 |  | 0 |
  Antigen A3-7, wk 19: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen A3-7, wk 19 | 0 |  |  |
  Antigen B8-1, wk 19: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-1, wk 19 | 0.32 |  |  |
  Antigen B8-3, wk 19: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-3, wk 19 | 0.99 |  |  |
  Antigen B8-4, wk 19: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-4, wk 19 | 0 |  |  |
  Antigen B8-5, wk 19: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-5, wk 19 | 0 |  |  |
  Antigen A3-1, wk 21: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-1, wk 21 | 0 |  | 0 |
  Antigen A3-2, wk 21: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-2, wk 21 | 0 |  | 0 |
  Antigen A3-3, wk 21: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-3, wk 21 | 0 |  | 0 |
  Antigen A3-4, wk 21: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-4, wk 21 | 0 |  | 0 |
  Antigen A3-5, wk 21: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-5, wk 21 | 0 |  | 0 |
  Antigen A3-6, wk 21: number analyzed (Participants) | 1 | 0 | 1 | 0
  Antigen A3-6, wk 21 | 0 |  | 0 |
  Antigen A3-7, wk 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen A3-7, wk 21 | 0 |  |  |
  Antigen B8-1, wk 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-1, wk 21 | 1.4 |  |  |
  Antigen B8-3, wk 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-3, wk 21 | 0.16 |  |  |
  Antigen B8-4, wk 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-4, wk 21 | 0 |  |  |
  Antigen B8-5, wk 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Antigen B8-5, wk 21 | 0 |  |  |
  Antigen B15-1, screening: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-1, screening |  | 0 |  |
  Antigen B15-2, screening: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-2, screening |  | 0 |  |
  Antigen B15-3, screening: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-3, screening |  | 0 |  |
  Antigen B15-4, screening: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-4, screening |  | 0 |  |
  Antigen B15-5, screening: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-5, screening |  | 0 |  |
  Antigen B44-1, screening: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B44-1, screening |  | 0 |  |
  Antigen A31-1, screening: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-1, screening |  | 0 |  |
  Antigen A31-2, screening: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-2, screening |  | 0 |  |
  Antigen B15-1, day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-1, day 1 |  | 0 |  |
  Antigen B15-2, day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-2, day 1 |  | 0 |  |
  Antigen B15-3, day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-3, day 1 |  | 0 |  |
  Antigen B15-4, day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-4, day 1 |  | 0 |  |
  Antigen B15-5, day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-5, day 1 |  | 0 |  |
  Antigen B44-1, day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B44-1, day 1 |  | 0 |  |
  Antigen A31-1, day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-1, day 1 |  | 0 |  |
  Antigen A31-2, day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-2, day 1 |  | 0 |  |
  Antigen B15-1, wk 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-1, wk 14 |  | 0 |  |
  Antigen B15-2, wk 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-2, wk 14 |  | 35 |  |
  Antigen B15-3, wk 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-3, wk 14 |  | 27.2 |  |
  Antigen B15-4, wk 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-4, wk 14 |  | 0 |  |
  Antigen B15-5, wk 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-5, wk 14 |  | 36.5 |  |
  Antigen B44-1, wk 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B44-1, wk 14 |  | 22.7 |  |
  Antigen A31-1, wk 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-1, wk 14 |  | 0 |  |
  Antigen A31-2, wk 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-2, wk 14 |  | 0 |  |
  Antigen B15-1, wk 17: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-1, wk 17 |  | 0 |  |
  Antigen B15-2, wk 17: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen B15-3, wk 17: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen B15-4, wk 17: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen B15-5, wk 17: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen B44-1, wk 17: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen A31-1, wk 17: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-1, wk 17 |  | 0 |  |
  Antigen A31-2, wk 17: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-2, wk 17 |  | 0 |  |
  Antigen B15-1, wk 19: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-1, wk 19 |  | 0 |  |
  Antigen B15-2, wk 19: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen B15-3, wk 19: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen B15-4, wk 19: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen B15-5, wk 19: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen B44-1, wk 19: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen A31-1, wk 19: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-1, wk 19 |  | 0 |  |
  Antigen A31-2, wk 19: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-2, wk 19 |  | 0 |  |
  Antigen B15-1, wk 21: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-1, wk 21 |  | 0 |  |
  Antigen B15-2, wk 21: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-2, wk 21 |  | 34.7 |  |
  Antigen B15-3, wk 21: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-3, wk 21 |  | 27.7 |  |
  Antigen B15-4, wk 21: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-4, wk 21 |  | 0 |  |
  Antigen B15-5, wk 21: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B15-5, wk 21 |  | 33.9 |  |
  Antigen B44-1, wk 21: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen B44-1, wk 21 |  | 17.4 |  |
  Antigen A31-1, wk 21: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-1, wk 21 |  | 0 |  |
  Antigen A31-2, wk 21: number analyzed (Participants) | 0 | 1 | 0 | 0
  Antigen A31-2, wk 21 |  | 0 |  |
  Antigen A3-8, screening: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-8, screening |  |  | 0 | 0
  Antigen A3-9, screening: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-9, screening |  |  | 0 | 0
  Antigen A3-10, screening: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-10, screening |  |  | 0 | 0
  Antigen A3-11, screening: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-11, screening |  |  | 0 | 0
  Antigen A3-8, day 1: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-8, day 1 |  |  | 0 | 0
  Antigen A3-9, day 1: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-9, day 1 |  |  | 0 | 0
  Antigen A3-10, day 1: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-10, day 1 |  |  | 0 | 0
  Antigen A3-11, day 1: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-11, day 1 |  |  | 0 | 0
  Antigen A3-8, wk 14: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-8, wk 14 |  |  | 0 | 1.15
  Antigen A3-9, wk 14: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-9, wk 14 |  |  | 0 | 1.08
  Antigen A3-10, wk 14: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-10, wk 14 |  |  | 0 | 0.9
  Antigen A3-11, wk 14: number analyzed (Participants) | 0 | 0 | 1 | 1
  Antigen A3-11, wk 14 |  |  | 10.8 | 0.14
  Antigen A3-8, wk 17: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-8, wk 17 |  |  | 0 |
  0Antigen A3-9, wk 17: number analyzed (Participants) | 0 | 0 | 1 | 0
  0Antigen A3-9, wk 17 |  |  | 0 |
  Antigen A3-10, wk 17: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-10, wk 17 |  |  | 0 |
  Antigen A3-11, wk 17: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-11, wk 17 |  |  | 0 |
  Antigen A3-8, wk 19: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-8, wk 19 |  |  | 0 |
  Antigen A3-9, wk 19: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-9, wk 19 |  |  | 0 |
  Antigen A3-10, wk 19: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-10, wk 19 |  |  | 0 |
  Antigen A3-11, wk 19: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-11, wk 19 |  |  | 0 |
  Antigen A3-8, wk 21: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-8, wk 21 |  |  | 0 |
  Antigen A3-9, wk 21: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-9, wk 21 |  |  | 0 |
  Antigen A3-10, wk 21: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-10, wk 21 |  |  | 0 |
  Antigen A3-11, wk 21: number analyzed (Participants) | 0 | 0 | 1 | 0
  Antigen A3-11, wk 21 |  |  | 0 |
  Antigen A3-12, screening: number analyzed (Participants) | 0 | 0 | 0 | 1
  Antigen A3-12, screening |  |  |  | 0
  Antigen A3-13, screening: number analyzed (Participants) | 0 | 0 | 0 | 1
  Antigen A3-13, screening |  |  |  | 0
  Antigen A3-12, day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Antigen A3-12, day 1 |  |  |  | 0
  Antigen A3-13, day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Antigen A3-13, day 1 |  |  |  | 0
  Antigen A3-12, wk 14: number analyzed (Participants) | 0 | 0 | 0 | 1
  Antigen A3-12, wk 14 |  |  |  | 0
  Antigen A3-13, wk 14: number analyzed (Participants) | 0 | 0 | 0 | 1
  Antigen A3-13, wk 14 |  |  |  | 1.48
  Antigen A3-12, wk 17: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen A3-13, wk 17: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen A3-12, wk 19: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen A3-13, wk 19: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen A3-12, wk 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  Antigen A3-13, wk 21: number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Safety and Tolerability of the Mature Dendritic Cell Vaccine (mDC3/8 Vaccines).
Description: Safety endpoint is type and number of adverse events. Tolerability endpoint is subject's completion or withdrawal from study treatment.
Time Frame: End of Study visit (10-28 days after last DC vaccine)
Population: Safety component is entered in the Adverse Events section.
Measure: Count of Participants; unit: Participants
Arm/Group | Mature Dendritic Cell (DC) Vaccine
Number analyzed (Participants) | 5
Participants
  Completed primary follow-up | 3
  Did not complete primary follow-up | 2

3. Secondary Outcome: Clinical Response to the mDC3/8 Vaccine(s)
Description: using RECIST 1.1
Time Frame: At the End of Study Treatment visit (~10-28 Days after the last DC vaccine)
Measure: Count of Participants; unit: Participants
Arm/Group | Mature Dendritic Cell (DC) Vaccine
Number analyzed (Participants) | 5
Participants
  Progressive disease | 2
  Not evaluable | 3

4. Secondary Outcome: Time to Progression Post-mDC3/8 Vaccine Administration
Description: based on RECIST 1.1 criteria, until occurrence of a censoring event
Time Frame: Up to 30 weeks after the first mDC3/8 Vaccine
Population: Results are presented per subject.
Measure: Number; unit: days
Arm/Group | Mature Dendritic Cell (DC) Vaccine
Number analyzed (Participants) | 5
days
  Subject 1: number analyzed (Participants) | 1
  Subject 1 | 113
  Subject 2: number analyzed (Participants) | 1
  Subject 2 | NA — Subject not evaluable.
  Subject 3: number analyzed (Participants) | 1
  Subject 3 | NA — Subject not evaluable.
  Subject 4: number analyzed (Participants) | 1
  Subject 4 | NA — Subject not evaluable.
  Subject 5: number analyzed (Participants) | 1
  Subject 5 | 80

5. Secondary Outcome: Safety and Side Effect Profile of the Dendritic Cell Vaccine (mDC3/8 Vaccines) Administered to Patients Given After a Single Dose of Cyclophosphamide.
Description: Assessed through collection of Adverse Events.
Time Frame: End of Study visit (10-28 days after last DC vaccine)
Population: These outcome measures are entered in the Adverse Events section.
Measure: Count of Participants; unit: Participants
Arm/Group | Mature Dendritic Cell (DC) Vaccine
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: Collection of AEs will begin at the time of the first apheresis procedure (Apheresis #1) and continue until subject discontinuation or the End of Study Visit. (week 30).
Arm/Group | Mature Dendritic Cell (DC) Vaccine
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mature Dendritic Cell (DC) Vaccine (N=5)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Surgical and medical procedures - Other (Palliative mass resection) (Surgical and medical procedures) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mature Dendritic Cell (DC) Vaccine (N=5)
Cardiac disorders - other )tachycardia) (Cardiac disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Toothache (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 2 (7)
Fatigue (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (3)
Parethesia (Nervous system disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03092453/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03092453/ICF_001.pdf